CLINICAL TRIAL: NCT03503552
Title: Body Composition and Risk for Development of Pre-diabetes in Post-menopausal Chinese Women in Singapore
Status: Completed | Type: Observational
Sponsor: JeyaKumar Henry (Other Government)
Collaborators: University of Auckland, New Zealand (Other); Massey University (Other); Institute of Materials Research and Engineering (IMRE) (Unknown)
Responsible Party: Sponsor-Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Organization: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Other Study IDs: 2014/01066
Record Dates: First submitted 2018-03-26; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Osteoporosis; Metabolic Syndrome
MeSH Terms: conditions — Osteoporosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to ascertain that novel imaging and metabolic markers can be used to identify as well as to validate and improve the detection of Singapore-Chinese women at increased risk of diabetes.

DETAILED DESCRIPTION:
Disproportionate non-communicable disease risk present in some ethnicities has been demonstrated and is amplified by increased weight gain. Relative to Malay and Caucasian populations, the prevalence of obesity increased sharply in people of Chinese and Indian ethnicity and diabetes risk is prevalent at a BMI of 21 (equivalent to a BMI >25 in Caucasian populations). It was also speculated that Chinese Singaporean women are prone to metabolic syndrome at a lower BMI. This study will recruit two groups of postmenopausal women with different BMI's and to measure markers for metabolic syndrome. These participants will visit Clinical Nutrition Research Centre for a single session and will undergo a whole body scan and a regional scan of the lumbar spine and femoral neck with a bone densitometer and fasting baseline blood and urine samples collected. Dual Energy X-ray Absorptiometry (DEXA) scan will provide percentage fat mass, fat in gram, whole body bone mineral content and total body lean mass. From these, gynoid and android fat distribution will be derived and appendicular lean mass will be calculated and an index calculated using kg/m2 to give an indication of relative muscle mass. In addition blood and urine samples will be collected for metabolic risk analysis. Participants will be also be undergoing a Quantitative Computed Tomography (QCT) scan which will allow true volumetric measurements of the lumbar spine and proximal femur independent of the body size. Volumetric density values will be measured in Hounsfield units transformed into Bone Mineral Density measurements using a calibration phantom underneath the patient. Magnetic Resonance Imaging of the 3rd lumbar vertebra and the right hip will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese women
* Aged 55 to 70 years
* Be 5 years past menopause
* Have not been diagnosed with type 1 diabetes

Exclusion Criteria:

* Have been diagnosed with Hyper or Hypo-thyroidism, Parathyroid disease, Diabetes Mellitus, Cushing's syndrome.
* Have Cancers
* Have Systemic Lupus Erythematosus and Rheumatoid Arthritis
* Respiratory Disease
* Had Operations such as Gastrectomy and Intestinal resection
* Have Liver Disease such as Liver cirrhosis
* On prescribed medication known to affect the study outcomes.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only post menopausal women
Study Population: Post menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 hour
  Measured using Air Displacement Plethysmograph (BOD POD)
Body composition | 1 hour
  Measured using Dual Energy X-Ray Absorptiometry
Body composition | 1 hour
  Measured using Magnetic Resonance Imaging (MRI)
Bone mineral density | Half an hour
  Measured using Dual Energy X-Ray Absorptiometry (DEXA)
Bone mineral density | Half an hour
  Measured using Quantitative Computed Tomography
Bone mineral density | Half an hour
  Measured using Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Blood biomarkers | Half an hour
  Measure of fasting blood glucose
Blood biomarkers | Half an hour
  Measure of fasting blood insulin
Blood biomarkers | Half an hour
  Measure of fasting blood lipid profile
Blood biomarkers | Half an hour
  Measure of fasting apolipoprotein A1
Blood biomarkers | Half an hour
  Measure of fasting apolipoprotein B
Blood biomarkers | Half an hour
  Measure of folate
Blood biomarkers | Half an hour
  Measure of vitamin B12
Blood biomarkers | Half an hour
  Measure of high-sensitive C-reactive protein
Blood biomarkers | Half an hour
  Measure of Parathyroid hormone
Urine Markers | Half an hour
  Measure urinary C-telopeptide of type II collagen

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No